CLINICAL TRIAL: NCT02762604
Title: Motor Imagery Intervention for Improving Gait and Cognition in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-3633; K01AG049829 (NIH); KL2TR001071 (NIH)
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imagined Gait Intervention (Experimental): During the phone-based imagined gait intervention, participants will be called by the experimenter three times a week and be asked to imagine walking, imagine talking and imagine walking-while-talking. They will also be asked to rate their visual and kinesthetic qualities of their images on a 1-5 scale following each trial.
  Interventions: Behavioral: Imagined Gait Intervention
- Visual Imagery Intervention (Active Comparator): During the phone-based visual imagery intervention, participants will be called three times a week by the experimenter and be asked to imagine concrete objects (e.g. octopus, teapot, and shovel). They will also be asked to rate their visual qualities of their images on a 1-5 scale following each trial.
  Interventions: Behavioral: Visual Imagery Intervention

INTERVENTIONS:
Behavioral: Imagined Gait Intervention — Phone-based imagined gait intervention: participants will be called by the experimenter three times a week and be asked to imagine walking, imagine talking and imagine walking-while-talking. They will also be asked to rate their visual and kinesthetic qualities of their images on a 1-5 scale following each trial.
  Arms: Imagined Gait Intervention
Behavioral: Visual Imagery Intervention — Phone-based visual imagery intervention: participants will be called three times a week by the experimenter and be asked to imagine concrete objects (e.g. octopus, teapot, and shovel). They will also be asked to rate their visual qualities of their images on a 1-5 scale following each trial.
  Arms: Visual Imagery Intervention

SUMMARY:
The investigators propose a single-blind randomized clinical trial to determine if seniors show improved mobility (walking speed) and cognition following motor imagery (imagined walking) training. They hypothesize that imagined walking can be used as a rehabilitative tool for improving walking speed and cognition in the elderly, because it engages and strengthens similar neural systems as actual walking and cognition.

DETAILED DESCRIPTION:
The proposed research aims to establish the efficacy of an imagined gait protocol for improving gait and cognition in the elderly. This imagined gait protocol involves imagined gait in single (imagined walking; iW) and dual-task (imagined walking while talking; iWWT) situations. A single-blind randomized clinical trial of 58 cognitively-healthy elderly with pre-post measures of gait, cognition, and functional Magnetic Resonance Imaging (fMRI) during imagined gait is proposed. The overall hypothesis is that imagined gait can be used as a rehabilitative tool for improving gait and cognition in the elderly because it engages and strengthens similar neural systems as actual gait and cognition. The first aim of this study is to establish the efficacy of our imagined gait protocol to improve gait and cognition in the elderly. We predict that our imagined gait intervention will improve gait velocity during actual walking and walking-while-talking conditions to a greater extent than the active control (visual imagery) intervention. We also predict that our imagined gait intervention will cognitive performance during dual-task walking conditions. The second aim of this study is to determine neuroplasticity changes in response to our imagined gait protocol. We predict that the neural systems engaged during imagined gait will change following our imagined gait intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 65 and 85 years and older, residing in the community.
* Able to speak English at a level sufficient to undergo study procedures.
* Plan to be in the area for the next 3 months.

Exclusion Criteria:

* Presence of dementia (telephone-based memory impairment screen < 5 or Ascertain Dementia 8-item Informant Questionnaire score > 1)
* Presence of gait disorder diagnosed by clinician (e.g. neuropathy).
* Any medical condition or chronic medication use (e.g. neuroleptics) that will compromise safety or affect cognitive functioning.
* Terminal illness with life expectancy <12 months.
* Progressive, degenerative neurologic disease (e.g. Parkinson's disease, ALS).
* Major psychiatric disorders such as Schizophrenia.
* Pacemaker or any permanent metal implants like hip prosthesis (other than tooth fillings) and claustrophobia.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena M Blumen, Ph.D, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blumen HM, Verghese J. Motor imagery of walking and walking while talking: a pilot randomized-controlled trial protocol for older adults. Neurodegener Dis Manag. 2017 Dec;7(6):353-363. doi: 10.2217/nmt-2017-0024. Epub 2017 Nov 22. PMID 29165011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization goal was 48 but two extra randomization slots were added as a buffer. Once 24 in each condition had been randomized, recruitment stopped, resulting in a total of 49 randomized participants.
Period: Overall Study
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Started | 25 | 24
Completed | 22 | 14
Not Completed | 3 | 10
Not completed — Lost to Follow-up | 2 | 7
Not completed — Study Suspension due to COVID pandemic | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.92 (5.28) | 72.79 (4.84) | 72.86 (5.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 17 | 15 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 6 | 16
  White | 10 | 12 | 22
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49
Years of Education [Mean (Standard Deviation); unit: years] — Population: Years of education for one participant in the Visual Imagery (VI) Intervention condition was missing
  years
    number analyzed (Participants) | 25 | 23 | 48
    (all) | 15.60 (3.06) | 16.52 (2.95) | 16.04 (3.01)

OUTCOME MEASURES:

1. Primary Outcome: Change in Walking Speed During Single and Dual-task Walking Conditions
Description: Change in gait speed (centimeters per second) measured during normal pace walking and walking while talking conditions using an instrumented pathway. A positive mean value is indicative of an improvement (increase) in gait speed post-intervention, whereas a negative mean value is indicative of a decrease in gait speed post-intervention.
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure).
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 25 | 10
centimeters per second
  Gait speed (normal pace) | -3.33 (14.13) | -0.53 (25.77)
  Gait speed (walking-while-talking) | 5.89 (20.44) | -10.55 (15.68)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in normal pace gait speed pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = -2.12, 95% CI 2-sided [-19.36 to 15.12], Standard Error of Mean 8.79 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups
Statistical Analysis 2: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in gait speed during walking while talking pre and post intervention; Test type: Superiority; Mean Difference (Net) = 17.19, 95% CI 2-sided [1.40 to 32.97], Standard Error of Mean 8.05 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

2. Secondary Outcome: Change in Cognitive Performance During Walking While Talking
Description: Change in cognitive performance was assessed by the number of correct letters/time (in seconds) generated during walking while talking (WWT). This exercise consists of having the participant walk around a computerized walkway while reciting alternate letters of the alphabet (WWT), starting with the letter "B." A positive mean value reflects an improvement in cognitive performance (increase in the number of correct letters/time generated) post-intervention; whereas, a negative mean value reflects worsening in cognitive performance (decrease in the number of correct letters/time generated) post-intervention.
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure). Data was also unable to be analyzed for 2 participants in the Visual Imagery group and 7 participants in the Imagined Gait group due to missing data.
Measure: Mean (Standard Deviation); unit: correct letters/second
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 18 | 8
correct letters/second | 0.19 (1.46) | -1.54 (1.50)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in correct letters generated pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 1.60, 95% CI 2-sided [0.21 to 2.99], Standard Error of Mean 0.71 — The estimate parameter reflects change in the number of correct letters generated pre to post intervention as a function intervention (Imagined Gait vs. Visual Imagery)

3. Secondary Outcome: Change in Blood-oxygen-level-dependent (BOLD) Signal During Dual-task Imagined Walking While Talking (iWWT) Conditions
Description: Change in blood-oxygen-level-dependent (BOLD) signal (neuroplasticity) during imagined walking and walking while talking (iWWT) conditions were measured using functional magnetic resonance imaging (fMRI). The mean values reported are changes in factor scores that reflect the overall change in BOLD signal pre- to post-intervention. Positive values reflect an increase in BOLD signal post-intervention, whereas, negative mean values reflect a decrease in BOLD signal post intervention. There are no minimum or maximum values or ranges or thresholds associated with the BOLD measure.
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure). Data was also unable to be analyzed for 2 participants in the Visual Imagery group and 2 participants in the Imagined Gait group due to incomplete tasks/sessions or corrupted data files.
Measure: Mean (Standard Deviation); unit: Factor score for BOLD signal
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 23 | 8
Factor score for BOLD signal | -2.98 (19.35) | -3.07 (11.89)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; Linear mixed effects model were used to compare changes in the functional activation/deactivation pattern (factor score) during imagery of walking-while talking (relative to walking and talking alone) pre and post intervention - as a function of of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 2.40, 95% CI 2-sided [-12.04 to 16.85], Standard Error of Mean 7.37 — The estimate parameter reflects change in functional activation/deactivation pattern from pre to post intervention as a function intervention (Imagined Gait vs. Visual Imagery)

4. Secondary Outcome: Change in Trail Making Test Form A
Description: Change in Trail Making Test Form A (TMT-A), is a timed measurement of attention and processing speed. Scoring is based on the time required to complete the task (i.e., drawing a line between 24 consecutive circles randomly arranged on a page) and ranges from 0-300 seconds with shorter time indicating better performance. A negative mean difference reflects an improvement pre to post intervention. The TMT-A uses all numbers (no letters) and includes correction of errors prompted by the examiner.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 25 | 10
seconds | -0.72 (19.16) | -1.45 (5.93)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; Linear mixed effects model were used to compare changes in trails a time pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = -0.54, 95% CI 2-sided [-14.15 to 13.07], Standard Error of Mean 6.94 — The estimate parameter is the difference in change pre to post intervention between Imagined Gait and Visual Imagery group

5. Secondary Outcome: Change in Trail Making Test Form B
Description: Change in Trail Making Test, Form B (TMT-B), is a timed measurement of attention, processing speed, and set-shifting. Scoring is based on the time required to complete the task (i.e., drawing a line between 24 consecutive circles randomly arranged on a page) and ranges from 0-300 seconds with shorter times indicating better performance. A negative mean difference reflects an improvement pre to post intervention. The TMT-B alternates between numbers and letters requiring the participant to switch between numbers and letters in consecutive order and includes correction of errors prompted by the examiner.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 25 | 10
seconds | 4.49 (54.18) | -9.54 (19.74)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; Linear mixed effects model were used to compare changes in trails b time pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = -12.21, 95% CI 2-sided [-51.92 to 27.51], Standard Error of Mean 20.26 — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Change in Trail Making Test Form B Minus Form A
Description: Change in Trail Making Test Form B (TMT-B) minus Form A (TMT-A), a timed measure of set-shifting. Scoring is based on the change in time between completing Form B compared to Form A. A negative mean difference reflects an improvement post intervention.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 25 | 10
seconds | 5.22 (50.28) | -8.09 (23.09)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; Linear mixed effects model were used to compare changes in trails B minus A time pre and post intervention; Test type: Superiority; Mean Difference (Net) = -10.83, 95% CI 2-sided [-48.12 to 26.47], Standard Error of Mean 19.03 — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Change in Letter Number Sequencing Task Score
Description: Change in scoring in the letter number sequencing task, a measure of item manipulation, was derived from the letter number sequencing subtest of the working memory domain within the Wechsler Adult Intelligence Scale (WAIS) III battery, a widely used intelligence test for adults. Scoring is based on the number of correctly sequenced letters and numbers with increasing (positive) mean scores indicating an improvement in task performance post intervention. A negative mean score reflects a decrease in task performance post intervention.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Correct sequences
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 25 | 10
Correct sequences | -0.55 (2.15) | 0.61 (1.84)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in correct letter number sequences pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = -0.93, 95% CI 2-sided [-2.65 to 0.79], Standard Error of Mean 0.88 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

8. Secondary Outcome: Change in Stroop Interference Test: Color-Word Minus Color Score
Description: Change in Stroop Interference Test: Color-Word (incongruent trials) minus Color (congruent trials) scores were determined. It is a measure of response competition and interference. Scoring is based on the time it takes to read (complete) incongruent trials relative to congruent trials. A negative mean value reflects an improvement in performance after the intervention. A positive mean value reflects an decrease in performance after the intervention.
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure) and for 1 participant in the Imagined Gait group due to missing data.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 24 | 10
seconds | -8.38 (30.14) | -14.47 (31.37)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in Stroop interference pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 1.39, 95% CI 2-sided [-24.00 to 26.78], Standard Error of Mean 12.95 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

9. Secondary Outcome: Change in Flanker Interference Task
Description: Change in the Flanker Interference Task measures how much interference is generated by the presentation of adjacent incongruent and congruent visual information. Scoring is based on the difference in reaction time (in milliseconds) between incongruent and congruent trials responded to correctly. A negative mean is indicative of improved interference post intervention and a positive mean value is indicative of worsening interference post intervention.
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure). Data was also unable to be analyzed for 7 participants in the Visual Imagery Group and 13 participants in the Imagined Gait group due to incomplete tasks/sessions or corrupted data files.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 12 | 3
milliseconds | -49.55 (108.85) | -94.69 (93.97)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in flanker interference pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 6.76, 95% CI 2-sided [-149.94 to 163.47], Standard Error of Mean 79.95 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

10. Secondary Outcome: Change in Stride Length
Description: Change in stride length were collected during walking while talking (WWT) conditions on an instrumented walkway. Stride length was defined as the distance between the heel points of 2 consecutive footfalls of the same foot and measured in centimeters (cm).
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure). Data was also unable to be analyzed for 1 participant in the Visual Imagery group and 6 participants in the Imagined Gait group due to missing data or corrupted data files.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 19 | 9
centimeters | 3.08 (9.33) | -11.49 (13.37)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in stride length during walking while talking pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 15.20, 95% CI 2-sided [5.99 to 24.41], Standard Error of Mean 4.70 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

11. Secondary Outcome: Change in Gait Variability
Description: Change in gait variability is collected during walking while talking on an instrumented walkway. Gait variability, defined as the stride-to-stride fluctuations in walking, was measured by the coefficient of variation (CV) of the mean value of stride-to stride time. CV reflects the level of gait rhythmicity, with lower values indicating greater rhythmicity. A negative mean CV reflects improved (less) variability post intervention whereas a positive mean CV value reflects worse (increased) variability. Stride time CV is closely associated with falls
Time Frame: Baseline and 3 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Coefficient of Variation (CV)
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 19 | 9
Coefficient of Variation (CV) | -0.17 (2.45) | 1.81 (1.56)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in gait variability during walking while talking pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = -1.96, 95% CI 2-sided [-3.73 to -0.20], Standard Error of Mean 0.90 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

12. Secondary Outcome: Change in Gait Domains
Description: Change in gait domains (summary measures reported in standard deviation units) derived from factor analysis of quantitative gait variables collected on an instrumented walkway during normal pace walking and walking while talking. Gait domain score is calculated by summing ratings for individual items and dividing by the maximum possible score for the domain, then multiplying by 100. The domain score ranges from 0 to 100, with higher scores reflecting more gait disturbance and lower scores reflecting less gait disturbance.
Time Frame: Baseline and 3 months
Population: Data were unable to be accurately computed for Gait Domain outcome measure due to incomplete data collection of the individual gait variable measurements which would have been summed to generate a Gait Domain Score. Since there was not enough data overall for the models to converge Gait Domain data was not able to be collected.
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Change in Free Cued Serial Recall Test
Description: Changes in free recall performance were based on the free cued serial recall test, a measure of verbal learning and memory. Scores range from 0 to 48. Mean values reflect the change in the number of items recalled pre and post intervention. A positive mean value indicates improved recall performance post intervention whereas a negative mean value reflects decreased performance post intervention.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: correct items recalled
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 25 | 10
correct items recalled | 1.14 (13.01) | -1.02 (5.81)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in total free recall pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 2.43, 95% CI 2-sided [-5.98 to 10.84], Standard Error of Mean 4.29 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

14. Other Pre Specified Outcome: Change in Delayed Figure Copy Recall on Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Description: Change in delayed figure copy recall performance from the RBANS assessment, a measure of spatial learning and memory. Figure copy recall scores range from 0 to 20. A positive mean is indicative of an increase in recall post intervention whereas a negative mean is indicative of a decrease in recall post intervention.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: correct items recalled
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 25 | 10
correct items recalled | 0.84 (5.83) | 2.47 (5.48)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in delayed figure copy recall pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = -1.94, 95% CI 2-sided [-5.88 to 2.00], Standard Error of Mean 2.01 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

15. Other Pre Specified Outcome: Change in Controlled Oral Word Fluency Test
Description: Change in the number of correct words generated on the controlled oral word fluency test, a measure of language processing. Scores range from 0 to 36. A positive mean reflects an improvement in language processing post intervention whereas a negative mean reflects worsening of language processing post intervention
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: correct items generated
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 25 | 10
correct items generated | 0.32 (18.37) | 2.90 (11.72)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in word fluency pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = -6.36, 95% CI 2-sided [-20.01 to 7.28], Standard Error of Mean 6.96 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

16. Other Pre Specified Outcome: Change in Semantic Fluency Test
Description: Change in the total number of correct words generated for each category on the semantic fluency test, a measure of language processing. Scores reflect the number of correct items generated in a 60 second window. A positive mean value reflects improved semantic fluency post intervention and a negative mean value reflects worsening of semantic fluency post intervention.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: correct words/minute
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 25 | 10
correct words/minute | 3.53 (17.04) | -4.20 (14.18)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in semantic fluency pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 5.73, 95% CI 2-sided [-6.51 to 17.97], Standard Error of Mean 6.25 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

17. Other Pre Specified Outcome: Change in Digit Symbol Substitution
Description: Change in number of correct digit symbols generated on the digit symbol substitution test (DSST), a measure of processing speed, attention and working memory. The number of correct symbols within the allowed time in seconds is measured. A positive mean reflects an improvement in the number of correct digit symbols generated post intervention whereas a negative mean value reflects fewer correct digits generated post intervention.
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Please note that data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure). Data was also unable to be analyzed for 1 participant in the Imagined Gait group due to missing data.
Measure: Mean (Standard Deviation); unit: correct digit symbols
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 24 | 10
correct digit symbols | 0.11 (20.10) | -2.61 (22.26)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in digit symbol substitution performance pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = -0.03, 95% CI 2-sided [-16.10 to 16.03], Standard Error of Mean 8.20; The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

18. Other Pre Specified Outcome: Modified Short Physical Performance Battery (SPPB) at Baseline
Description: SPPB is a measure of lower extremity function and includes a balance test, a chair stand test and a gait speed test. Because gait speed/velocity was our primary outcome, only administered the balance and chair stand tests were administered. Thus, possible scores range from 0-8 (rather than the typical 0-12) with 0 being worst performance and 8 being best performance.
Time Frame: Baseline
Population: SPPB was only administered at baseline (only the balance and chair tests were administered). Change analyses were not performed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 24 | 10
score on a scale | 6.79 (1.17) | 6.30 (1.34)

19. Other Pre Specified Outcome: Change in Immediate Maze Task Performance
Description: Change in mean immediate maze performance (time in seconds), a measure of spatial navigation and memory, were determined. A negative mean value represents an improvement in immediate maze performance post intervention whereas a positive mean value represents worsening of maze performance post intervention.
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure). Data was also unable to be analyzed for 5 participants in the in the Imagined Gait group due to missing data.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 20 | 10
seconds | 9.27 (23.21) | 4.09 (6.48)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in immediate maze performance pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 3.64, 95% CI 2-sided [-11.14 to 18.42], Standard Error of Mean 7.54 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

20. Other Pre Specified Outcome: Change in Delayed Maze Task Performance
Description: Change in mean delayed maze performance (time in seconds), a measurement of spatial navigation and memory, were determined. A negative mean value represents an improvement in delayed maze performance post intervention, whereas a positive mean performance time represents worsening delayed maze performance post intervention
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure). Data was also unable to be analyzed for 4 participants in the in the Imagined Gait group due to missing data.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 21 | 10
seconds | 7.25 (42.07) | 4.04 (5.23)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in delayed maze performance pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 3.26, 95% CI 2-sided [-20.65 to 27.18], Standard Error of Mean 12.20 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

21. Other Pre Specified Outcome: Change in Errors on Maze Task
Description: The number of errors during maze performance, a measure of spatial navigation and memory, will be assessed. A negative mean result is indicative of an improvement (fewer errors) post intervention whereas a positive mean result is indicative of a reduction in performance (more errors) post intervention.
Time Frame: Baseline and 3 months
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 20 | 10
errors | -0.27 (1.03) | 0.14 (0.32)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in maze errors pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 0.22, 95% CI 2-sided [-0.45 to 0.90], Standard Error of Mean 0.34 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

22. Other Pre Specified Outcome: Change in Geriatric Depression Scale
Description: The Geriatric Depression Scale (GDS) will be used to to determine mean changes in depressive symptoms from baseline. Scores range from 0 to 30. Scores of 0 - 9 are considered normal, 10 - 19 indicate mild depression and 20 30 indicate severe depression. As such, higher scores are indicative of more severe depressive symptoms. A positive mean value reflects an increase in depressive symptoms post-intervention whereas a negative value reflects a decrease in depressive symptoms post intervention.
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure). Data was also unable to be analyzed for 3 participants in the in the Imagined Gait group and 2 participants in the in the Visual Imagery group due to missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 22 | 8
score on a scale | 0.11 (2.30) | 0.00 (2.39)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in depressive symptoms pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 0.26, 95% CI 2-sided [-1.74 to 2.26], Standard Error of Mean 1.02 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

23. Other Pre Specified Outcome: Change in Beck Anxiety Inventory
Description: Change in symptoms of anxiety. Scores range from 0 to 84 with higher values reflecting more anxiety symptoms. A negative mean reflects a reduction in anxiety symptoms post intervention and a positive mean value reflects an increase in anxiety symptoms post intervention
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure). Data was also unable to be analyzed for 6 participants in the in the Imagined Gait group and 2 participants in the in the Visual Imagery group due to missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 19 | 8
score on a scale | 0.24 (1.92) | 1.00 (4.16)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in anxiety symptoms pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = -0.95, 95% CI 2-sided [-3.38 to 1.49], Standard Error of Mean 1.24 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

24. Other Pre Specified Outcome: Change in Gray Matter Cortical Thickness
Description: Change in mean Cortical Thickness obtained from T1-weighted structural images. A positive mean value reflects an increase in cortical thickness post intervention and a negative mean value reflects a decrease in cortical thickness post intervention
Time Frame: Baseline and 3 months
Population: Overall number of participants analyzed includes all randomized participants with baseline measures. Data was unable to be analyzed for 14 participants in the Visual Imagery group due to a protocol deviation (incorrect intervention procedure). Data was also unable to be analyzed for 2 participants in the in the Visual Imagery group due to missing data.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 25 | 8
millimeters | -0.03 (0.09) | -0.07 (0.03)
Statistical Analysis 1: Comparison: Imagined Gait Intervention vs Visual Imagery Intervention; A linear mixed effects model was used to compare changes in cortical thickness pre and post intervention - as a function of intervention (Imagined Gait vs. Visual Imagery); Test type: Superiority; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.04 to 0.12], Standard Error of Mean 0.04 — The estimate parameter reflects the difference in pre to post change between Imagined Gait and Visual Imagery groups

25. Other Pre Specified Outcome: Change in White Matter Integrity
Description: Change in White Matter Integrity obtained from diffusion-weighted imaging. Increased white matter integrity is associated with improved cognitive performance whereas decreased white matter integrity is associated with decreased cognitive performance.
Time Frame: Baseline and 3 months
Population: Results were unable to be computed for White Matter Integrity due to limited data.
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 0 | 0

26. Other Pre Specified Outcome: Change in White Matter Hyperintensities
Description: Change in White Matter Hyperintensities obtained from Fluid-Attenuated Inversion Recovery imaging. Increased white matter hyperintensities may be indicative of unfavorable outcomes.
Time Frame: Baseline and 3 months
Population: Results were unable to be computed for White Matter Hyperintensities due to limited data.
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Participants were queried weekly about falls and any changes to their health.
Arm/Group | Imagined Gait Intervention | Visual Imagery Intervention
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/24
Other Adverse Events (participants affected / at risk) | 5/25 | 11/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imagined Gait Intervention (N=25) | Visual Imagery Intervention (N=24)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Participant was recruited into the study 06/01/2021 and completed 21 intervention sessions prior to onset. Participant was diagnosed with pneumonia on 8/8/2021 and was hospitalized for treatment. Participant resumed intervention calls on 9/13/21
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imagined Gait Intervention (N=25) | Visual Imagery Intervention (N=24)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back/shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Pain in lower extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (4)
Pain in upper extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Enlarged prostate (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT02762604/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT02762604/ICF_001.pdf